CLINICAL TRIAL: NCT03332355
Title: (STM-03) Phase I Study of Procaspase Activating Compound-1 (PAC-1) in the Treatment of Advanced Malignancies - Component 2
Brief Title: Procaspase Activating Compound-1 (PAC-1) in the Treatment of Advanced Malignancies - Component 2
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Vanquish Oncology, Inc. (Industry)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0058
Record Dates: First submitted 2017-10-16; First posted 2017-11-06 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2022-06

CONDITIONS: Glioblastoma Multiforme; Anaplastic Astrocytoma
Keywords: glioblastoma multiforme; anaplastic astrocytoma; high grade glioma; temozolomide; PROCASPASE ACTIVATING COMPOUND-1 (PAC-1); advanced malignancy; maximal tolerated dose (MTD)
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Glioma | interventions — (4-benzylpiperazin-1-yl)acetic acid (3-allyl-2-hydroxybenzylidene)hydrazine

STUDY DESIGN:
Intervention Model Description: PAC-1 in combination with temozolomide (Component 2): after the MTD is established for single agent PAC-1 in Component 1, a modified-Fibonacci dose-escalation 3+3 design starts in Component 2, at a PAC-1 dose one level lower than the MTD of PAC-1 established in the single agent PAC-1 component (i.e., Component 1) and 150 mg/m2 dose of temozolomide given for the 5 days starting at day 8 of cycle 1 in cohorts of 3-6 patients. The combination cohort that reaches MTD will expanded to at least 9 patients, similar to the PAC-1 alone cohort at MTD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PAC-1 in combination with temozolomide (Experimental): Temozolomide (PO) will be dosed at 150 mg (adjusted for body size area [m2]) daily for 5 days starting on day 8 at cycle 1, and then for each successive cycle. In Component 2, the first PAC-1 dose will be 1 dose level lower than the PAC-1 MTD established in Component 1, and the maximum dose will not exceed 450 mg. PAC-1 will be taken in the morning on days 1-21 in each 28-day cycle.
  Interventions: Drug: PAC-1 Compound

INTERVENTIONS:
Drug: PAC-1 Compound — PAC-1 in combination with temozolomide (Component 2): after the MTD is established for single agent PAC-1 in Component 1, a modified-Fibonacci dose-escalation 3+3 design starts in Component 2, at a PAC-1 dose one level lower than the MTD of PAC-1 established in the single agent PAC-1 component (i.e., Component 1). PAC-1 will be taken in the morning on days 1-21 in each 28 day cycle. Temozolomide 150 mg/m2 dose is given for the 5 days starting at day 8 of cycle 1 in cohorts of 3-6 patients. The combination cohort that reaches MTD will expanded to at least 9 patients, similar to the PAC-1 alone cohort at MTD.
  Other Names: Temozolamide

SUMMARY:
The primary objectives of this study are to determine the maximal tolerated dose (MTD) of PAC-1 in combination with temozolomide in patients with high grade glioma: glioblastoma multiforme (GBM) or anaplastic astrocytoma after progression following standard first line therapy (Component 2), by evaluation of toxicity and tolerability.

DETAILED DESCRIPTION:
PAC-1 in combination with temozolomide (Component 2): after the MTD is established for single agent PAC-1 in Component 1, a modified-Fibonacci dose-escalation 3+3 design starts in Component 2, at a PAC-1 dose one level lower than the MTD of PAC-1 established in the single agent PAC-1 component (i.e., Component 1) and 150 mg/m2 dose of temozolomide given for the 5 days starting at day 8 of cycle 1 in cohorts of 3-6 patients. The combination cohort that reaches MTD will expanded to at least 9 patients, similar to the PAC-1 alone cohort at MTD. For all dose cohorts, pharmacokinetics of PAC-1 will be assessed following doses administered on days 1 and 11 of the first cycle. Temozolomide pharmacokinetics will be performed on Day 11 of the first cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age
2. Diagnosis of advanced solid tumor or hematologic malignancy (limited to lymphoma) that has failed or become intolerant to standard therapy (Component 1 - single agent PAC-1) Note: Gliomas are excluded from Component 1 (see exclusion #19)
3. Diagnosis of high grade glioma: glioblastoma multiforme (GBM) or anaplastic astrocytoma after progression following treatment with standard first line therapy (Component 2 - PAC-1 in combination with temozolomide).
4. Has measurable disease, defined as at least 1 tumor that fulfills the criteria for a target lesion according to RECIST 1.1 (Component 1).
5. For patients in study Component 2 measurable disease RANO criteria will be used.
6. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 (see Appendix 4)
7. Has adequate hepatic function defined as total bilirubin < 1.5 mg/dL, serum albumin > 3.0 gm/dL, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 1.5 × upper limit of normal (ULN) or < 3 x ULN for subjects with known hepatic metastases
8. Has adequate renal function defined as serum creatinine < 1.5 × ULN
9. Has adequate bone marrow function defined as a hemoglobin ≥ 10 g/dL, absolute neutrophil count (ANC) ≥ 1.5 × 109/L, and platelet count ≥ 100 × 109/L
10. Patients taking antiepileptic drugs (AED) must be on stable doses of AED for at least two weeks prior to registration and have no episode of seizures for at least 14 days prior to registration. Because some AEDs enhance or inhibit enzymes that may affect PAC-1 metabolism, those AEDs will not be permitted in this study. The AEDs that are and are not permissible are in Appendix 6.
11. Patient must be able to take oral medication and to maintain a fast as required for 2 hours before and 1 hour after capsule(s) administration
12. Must be willing and able to comply with study visits and procedures
13. Has read, understood and signed the informed consent form (ICF) approved by the Institutional Review Board/Independent Ethics Committee (IRB/IEC)
14. Women of childbearing potential (WOCP) must not be pregnant (confirmed by a negative pregnancy test, with a serum B-HCG with a sensitivity of 50 mL U/L within 7 days of study treatment) or breast-feeding. In addition, a medically acceptable method of birth control must be used such as an oral, implantable, injectable, or transdermal hormonal contraceptive, an intrauterine device (IUD), use of a double barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream), or total abstinence during the study participation and for one month after last dose of study drug(s). Women who are postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) are not considered to be WOCP.
15. Men who are not surgically or medically sterile must agree to use an acceptable method of contraception. Male patients with female sexual partners who are pregnant, possibly pregnant, or who could become pregnant during the study must agree to use condoms at least one month after the last dose of study drug. Total abstinence for the same study period is an acceptable alternative.
16. Prior systemic treatments for metastatic disease are permitted but may not be ongoing, including targeted therapies, biologic response modifiers, chemotherapy, hormonal therapy, or investigational therapy (see Exclusion #20).
17. Willingness to donate blood for biomarker studies related to the type of therapies used in this trial and the tumor types being treated

    Exclusion Criteria:
18. Had surgery within 4 weeks prior to study treatment except for minor procedures (hepatic biliary stent placement is allowed)
19. For Component 1 (PAC-1 alone), gliomas are excluded, as well as any history of brain metastases, seizures or underlying brain injury (e.g., traumatic brain injury, or hemorrhagic or ischemic stroke)
20. Patients may not have received cytotoxic chemotherapy, targeted therapies, biologic response modifiers, chemotherapy, and hormonal therapy within the last 3 weeks, or nitrosureas within the last 6 weeks prior to study treatment.
21. Has a known hypersensitivity to temozolomide (this criterion applies only in Component 2)
22. Has a history of blood clots, pulmonary embolism, or deep vein thrombosis unless controlled by anticoagulant treatment (patient must be on stable dose for 2 weeks)
23. Has a history of an arterial thromboembolic event within the prior six months including cerebrovascular accident, transient ischemic attack, myocardial infarction, or unstable angina.
24. Has uncontrolled human immunodeficiency virus (HIV) (defined as HIV RNA >500 copies/ml and CD4+ count<200/mm3 on antiretroviral therapy) infection or hepatitis B (defined as ALT > 1 x ULN, and HBV DNA >2000 IU/ml) or hepatitis C (defined as ALT > 1 x ULN, persistent viremia on antiviral therapy) infections.
25. Has any clinically significant infection, i.e., any acute viral, bacterial, or fungal infection that requires specific treatment (anti-infective treatment has to be completed ≥ 7 days prior to study entry)
26. Has any other severe, uncontrolled medical condition, including uncontrolled diabetes mellitus (defined as a Hemoglobin A1C≥ 9% in patients with a prior history of diabetes, 28 days prior to study ) or clinical signs of unstable congestive heart failure (Stage III-IV of the New York Heart Association Functional Classification) (Appendix 5).
27. Radiation therapy to more than 25% of the bone marrow. Whole pelvic radiation is considered to be over 25%.
28. Prior allogeneic bone marrow or organ transplantation.
29. > Grade 1 peripheral neuropathy within 14 days before enrollment.
30. Pregnant or breastfeeding - temozolomide is Pregnancy Category D - can cause fetal harm. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
31. Patient has received other investigational drugs within 14 days prior to study treatment.
32. Other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for enrollment in this study.
33. Abnormalities on 12-lead electrocardiogram (ECG) considered by the investigator to be clinically significant (such as acute ischemia, left bundle branch block, ventricular arrhythmias) or baseline prolongation of the rate-corrected QT interval (e.g., repeated demonstration of QTc interval > 480 milliseconds).
34. Presence of any non-healing wound, fracture, or ulcer within 28 days prior to the first dose of study drug.
35. Has any condition that, in the opinion of the investigator, might jeopardize the safety of the patient or interfere with protocol compliance
36. Has any mental or medical condition that prevents the patient from giving informed consent or participating in the trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | During treatment cycle 1 (first 28 days)
  MTD, defined as the highest tolerated dose of PAC-1 tested in combination with temozolomide in patients with high grade glioma.

SECONDARY OUTCOMES:
Adverse Effects | Up to 30 days post final dose
  Toxicity will be graded using the Common Terminology Criteria for Adverse Events version 4 (CTCAE v4)
Disease Response | Through study completion, an average of one year
  Disease response will be assessed by RANO criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Oana C Danciu, M.D., Principal Investigator — Unversity of Illinois at Chicago
Locations (3):
- United States (3):
  - University of Illinois at Chicago, Chicago, Illinois
  - Johns Hopkins Cancer Center, Baltimore, Maryland
  - Regions Hospital, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No